CLINICAL TRIAL: NCT04011969
Title: The Role of Gut Microbiome and Chronic Inflammation in Young-onset Colorectal Cancer: Next-generation Sequencing (NGS) as a Screening Method
Brief Title: The Role of Gut Microbiome and Chronic Inflammation in Young-onset Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Murdani Abdullah, Professor, Fakultas Kedokteran Universitas Indonesia
Other Study IDs: 19-05-0528
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Cancer
Keywords: chronic inflammation; young-onset colorectal cancer; gut microbiome; NGS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal cancer suspects: Patients suspected with colorectal cancer who come to our hospital to conduct colonoscopy procedure will be recruited for this study and will undergo a series of examinations.
  Interventions: Diagnostic Test: Score assessment; Diagnostic Test: Blood sampling; Diagnostic Test: Fecal sampling

INTERVENTIONS:
Diagnostic Test: Score assessment — Asia Pacific Colorectal Screening (APCS) is a validated tool to predict the risk of colorectal cancer in asymptomatic Asian population. The scoring system comprises of three categories: low risk (score 0-1), moderate risk (score 2-3) and high risk (score 4-7). Patients with moderate and high risk will undergo further examinations.
Diagnostic Test: Blood sampling — Blood samples will be taken before colonoscopy procedure to evaluate the level of serum CEA by ELISA method and to evaluate the presence of NF-ҡB by immunohistochemical method.
  1. Carcinoembryonic antigen (CEA) is a well-known marker for colorectal cancer. A pre-treatment serum CEA level of ≥ 5 ng/mL is associated with poor prognosis in colorectal cancer patients.
  2. NF-ҡB is a chronic inflammation marker found in colorectal cancer patients.
Diagnostic Test: Fecal sampling — Fecal samples will be taken before colonoscopy procedure to be tested for FIT and to evaluate the gut microbiome.
  1. Fecal immunochemical test (FIT) is a recommended screening method for colorectal cancer. Detection of hemoglobin over a certain level in fecal samples indicated a positive FIT. Patients with positive FIT will undergo further examinations.
  2. Gut microbiome examination will be conducted with next generation sequencing (NGS) method.

SUMMARY:
This study aims to investigate the role of gut microbiome pattern and inflammation marker NF-ҡB in young-onset colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 35 years old
2. Suspected with colorectal cancer and undergoing a colonoscopy procedure
3. No history of colorectal cancer treatment

Exclusion Criteria:

1. Unwilling to provide fecal and blood sample
2. Incomplete colonoscopy procedure due to any reasons

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suspected with colorectal cancer who come to our hospital to conduct colonoscopy procedure will be recruited for this study and will undergo a series of examinations. Since this is a pilot study to obtain gut microbiome pattern on colorectal cancer patients, the number of samples is determined by the researchers: 100 subjects for neoplasm and 50 subjects for non-neoplasm (according to histopathology report)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome | pre-colonoscopy, approximately 1 day before colonoscopy
  Gut microbiome examination will be conducted with next generation sequencing (NGS) method
Asia Pacific Colorectal Screening (APCS) score | pre-colonoscopy, approximately 1 day before colonoscopy
  Asia Pacific Colorectal Screening (APCS) is a validated tool to predict the risk of colorectal cancer in asymptomatic Asian population. The scoring system comprises of three categories: low risk (score 0-1), moderate risk (score 2-3) and high risk (score 4-7). Patients with moderate and high risk will undergo further examinations
Carcinoembryonic antigen (CEA) serum level | pre-colonoscopy, approximately 1 day before colonoscopy
  Carcinoembryonic antigen (CEA) is a well-known marker for colorectal cancer. A pre-treatment serum CEA level of ≥ 5 ng/mL is associated with poor prognosis in colorectal cancer patients.
Presence of NF-ҡB | pre-colonoscopy, approximately 1 day before colonoscopy
  NF-ҡB is a chronic inflammation marker found in colorectal cancer patients. Presence of NF-ҡB is assessed with immunohistochemical method. The result is considered positive if accumulated score ≥ 3.
Fecal immunochemical test (FIT) | pre-colonoscopy, approximately 1 day before colonoscopy
  Fecal immunochemical test (FIT) is a recommended screening method for colorectal cancer. Detection of hemoglobin over a certain level in fecal samples indicated a positive FIT. Patients with positive FIT will undergo further examinations

CONTACTS AND LOCATIONS:
Overall Officials: Murdani Abdullah, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- RSUPN dr. Cipto Mangunkusumo (Cipto Mangunkusumo Hospital), Jakarta, DKI Jakarta, Indonesia

DOCUMENTS (1):
  • Study Protocol (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT04011969/Prot_000.pdf